CLINICAL TRIAL: NCT01398696
Title: Impact of Four Patient Information Leaflets (PIL) on Patient Behaviour : a Randomised Controlled Trial in Primary Care.
Brief Title: Impact of Four Patient Information Leaflets (PIL) on Patient Behaviour
Acronym: PIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: n° IRB 5891
Record Dates: First submitted 2011-04-19; First posted 2011-07-20 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Gastroenteritis; Pharyngitis
Keywords: Patient Information Leaflets; primary care; patient behaviour; pharyngitis; gastroenteritis
MeSH Terms: conditions — Gastroenteritis; Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Information Leaflets (Active Comparator): Patient Information Leaflets (PIL) is given to the patient during consultation
  Interventions: Procedure: Patient Information Leaflets
- usual consultation without PIL (Placebo Comparator): no particular intervention during consultation for the patient.
  Interventions: Procedure: usual consultation

INTERVENTIONS:
Procedure: Patient Information Leaflets — Patient Information Leaflets (PIL) about adult gastroenteritis, children gastroenteritis, adult pharyngitis or either children pharyngitis in consultation room
  Arms: Patient Information Leaflets
Procedure: usual consultation — No particular intervention during consultation for the Patient. No Information Leaflets (PIL) is given
  Arms: usual consultation without PIL

SUMMARY:
To assess the impact of four Patient Information Leaflets (PIL) on patient behaviour in primary care.

DETAILED DESCRIPTION:
A patient who visited, for a gastroenteritis or a pharyngitis, one GP of the intervention group, received a Patient Information Leaflets (PIL) related to his disease and his age: either the gastroenteritis leaflet for adult or the one for child, either the pharyngitis leaflet for adult or the one for child.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient.
* Minor child accompanied by a responsible adult.
* The patient or the caregiver must be reachable by telephone within ten to fifteen days following the consultation.

Exclusion Criteria:

* Illiterate patient
* Patient refusing follow-up call.
* Patient with visual or hearing impairment.
* Patient non-Francophone.
* Private patient of liberty by judicial or administrative.
* Person being a measure of legal protection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was the mean behaviour score | In ten to fifteen days after patient after the visit
  All patients were called, ten to fifteen days after the visit, to answer a questionnaire on their behaviour related to the disease since they visited the GP. It permitted to calculate a behaviour score. Better was the score, better was the patient's behaviour related to his disease.

SECONDARY OUTCOMES:
the mean comprehension score | in ten to fifteen days after the visit
  All patients (or their parent) were called, ten to fifteen days after the visit, to answer a questionnaire on their comprehension related to the disease since they visited the GP. It permitted to calculate a comprehension score. Better was this score, better was the patient's comprehension.
number of visit of patient's family for the same pathology | in ten to fifteen days after the visit
  we get the information by a phone call to the patient, in ten to fifteen days after the visit

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Sustersic, GP, Study Director — University Hospital, Grenoble; Jean-Luc Bosson, PHD, Study Director — University Hospital, Grenoble; LUCILE REIN, MD, Principal Investigator — University Hospital, Grenoble; EVA JEANNET, MD, Principal Investigator — University Hospital, Grenoble
Locations (23):
- France (23):
  - General practitioner office, Beaulieu-sur-Mer
  - General practitioner office, Chambéry
  - General practitioner office, Charolles
  - General practitioner office, Chirens
  - General practitioner office, Coublevie
  - General practitioner office, Échirolles
  - General practitioner office, Grenoble
  - University Hospital Grenoble, Grenoble
  - General practitioner office, Juan-les-Pins
  - General practitioner office, La Buisse
  - General practitioner office, La Murette
  - General practitioner office, Le Plessis-Robinson
  - General practitioner office, Lyon
  - General practitioner office, Massy
  - General practitioner office, Megève
  - General practitioner office, Saint-Étienne-de-Crossey
  - General practitioner office, Saint-Marcellin
  - General practitioner office, Saint-Martin-d'Hères
  - General practitioner office, Saint-Priest
  - General practitioner office, Saint-Sorlin
  - General practitioner office, Ugine
  - General practitioner office, Valence
  - General practitioner office, Voiron

REFERENCES:
- [Background] Stewart M, Brown JB, Donner A, McWhinney IR, Oates J, Weston WW, Jordan J. The impact of patient-centered care on outcomes. J Fam Pract. 2000 Sep;49(9):796-804. PMID 11032203
- [Background] Kitching JB. Patient information leaflets--the state of the art. J R Soc Med. 1990 May;83(5):298-300. doi: 10.1177/014107689008300506. No abstract available. PMID 2380944
- [Background] Kenny T, Wilson RG, Purves IN, Clark J Sr, Newton LD, Newton DP, Moseley DV. A PIL for every ill? Patient information leaflets (PILs): a review of past, present and future use. Fam Pract. 1998 Oct;15(5):471-9. doi: 10.1093/fampra/15.5.471. PMID 9848435
- [Background] Little P, Griffin S, Kelly J, Dickson N, Sadler C. Effect of educational leaflets and questions on knowledge of contraception in women taking the combined contraceptive pill: randomised controlled trial. BMJ. 1998 Jun 27;316(7149):1948-52. doi: 10.1136/bmj.316.7149.1948. PMID 9641933
- [Background] Little P, Dorward M, Warner G, Moore M, Stephens K, Senior J, Kendrick T. Randomised controlled trial of effect of leaflets to empower patients in consultations in primary care. BMJ. 2004 Feb 21;328(7437):441. doi: 10.1136/bmj.37999.716157.44. Epub 2004 Feb 13. PMID 14966078
- [Background] Coudeyre E, Givron P, Vanbiervliet W, Benaim C, Herisson C, Pelissier J, Poiraudeau S. [The role of an information booklet or oral information about back pain in reducing disability and fear-avoidance beliefs among patients with subacute and chronic low back pain. A randomized controlled trial in a rehabilitation unit]. Ann Readapt Med Phys. 2006 Nov;49(8):600-8. doi: 10.1016/j.annrmp.2006.05.003. Epub 2006 May 26. French. PMID 16793163
- [Background] Coudeyre E, Poiraudeau S, Revel M, Kahan A, Drape JL, Ravaud P. Beneficial effects of information leaflets before spinal steroid injection. Joint Bone Spine. 2002 Dec;69(6):597-603. doi: 10.1016/s1297-319x(02)00457-8. PMID 12537268
- [Background] McIntosh A, Shaw CF. Barriers to patient information provision in primary care: patients' and general practitioners' experiences and expectations of information for low back pain. Health Expect. 2003 Mar;6(1):19-29. doi: 10.1046/j.1369-6513.2003.00197.x. PMID 12603625
- [Background] Watkins CJ, Papacosta AO, Chinn S, Martin J. A randomized controlled trial of an information booklet for hypertensive patients in general practice. J R Coll Gen Pract. 1987 Dec;37(305):548-50. PMID 3503941
- [Background] Roberts L, Little P, Chapman J, Cantrell T, Pickering R, Langridge J. The back home trial: general practitioner-supported leaflets may change back pain behavior. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1821-8. doi: 10.1097/00007632-200209010-00002. PMID 12221342
- [Background] Johnson LK, Edelman A, Jensen J. Patient satisfaction and the impact of written material about postpartum contraceptive decisions. Am J Obstet Gynecol. 2003 May;188(5):1202-4. doi: 10.1067/mob.2003.308. PMID 12748478
- [Background] Mancini J, Nogues C, Adenis C, Berthet P, Bonadona V, Chompret A, Coupier I, Eisinger F, Fricker JP, Gauthier-Villars M, Lasset C, Lortholary A, N'Guyen TD, Vennin P, Sobol H, Stoppa-Lyonnet D, Julian-Reynier C. Impact of an information booklet on satisfaction and decision-making about BRCA genetic testing. Eur J Cancer. 2006 May;42(7):871-81. doi: 10.1016/j.ejca.2005.10.029. Epub 2006 Mar 23. PMID 16563745
- [Background] Al-Asfour A, Andersson L. The effect of a leaflet given to parents for first aid measures after tooth avulsion. Dent Traumatol. 2008 Oct;24(5):515-21. doi: 10.1111/j.1600-9657.2008.00651.x. PMID 18821954
- [Background] Carre PC, Roche N, Neukirch F, Radeau T, Perez T, Terrioux P, Ostinelli J, Pouchain D, Huchon G. The effect of an information leaflet upon knowledge and awareness of COPD in potential sufferers. A randomized controlled study. Respiration. 2008;76(1):53-60. doi: 10.1159/000115947. Epub 2008 Feb 5. PMID 18253024
- [Background] Scala D, Cozzolino S, D'Amato G, Cocco G, Sena A, Martucci P, Ferraro E, Mancini AA. Sharing knowledge is the key to success in a patient-physician relationship: how to produce a patient information leaflet on COPD. Monaldi Arch Chest Dis. 2008 Jun;69(2):50-4. doi: 10.4081/monaldi.2008.395. PMID 18837416
- [Background] Vetto JT, Dubois PM, Vetto IP. The impact of distribution of a patient-education pamphlet in a multidisciplinary breast clinic. J Cancer Educ. 1996 Fall;11(3):148-52. doi: 10.1080/08858199609528418. PMID 8877574
- [Background] Leichtnam-Dugarin L, Carretier J, Delavigne V, Brusco S, Hoarau H, Philip T, Fervers B; Comite d'Organisation des Standards, Options et Recommentations SAVOIR; Federation Nationale des Centres de lutte contre le cancer; Ligue contre le Cancer; Federation Hospitaliere de France; Federation Nationale de Cancerologie des CHRU; Federation Francaise de Cancerologie. [The SOR SAVOIR Patient, a project of patient information and education]. Cancer Radiother. 2003 Jun;7(3):210-2. doi: 10.1016/s1278-3218(03)00037-4. No abstract available. French. PMID 12834779
- [Background] Roland M, Dixon M. Randomized controlled trial of an educational booklet for patients presenting with back pain in general practice. J R Coll Gen Pract. 1989 Jun;39(323):244-6. PMID 2556518
- [Background] Macfarlane JT, Holmes WF, Macfarlane RM. Reducing reconsultations for acute lower respiratory tract illness with an information leaflet: a randomized controlled study of patients in primary care. Br J Gen Pract. 1997 Nov;47(424):719-22. PMID 9519518
- [Background] Macfarlane J, Holmes W, Gard P, Thornhill D, Macfarlane R, Hubbard R. Reducing antibiotic use for acute bronchitis in primary care: blinded, randomised controlled trial of patient information leaflet. BMJ. 2002 Jan 12;324(7329):91-4. doi: 10.1136/bmj.324.7329.91. PMID 11786454
- [Background] Vuorma S, Rissanen P, Aalto AM, Hurskainen R, Kujansuu E, Teperi J. Impact of patient information booklet on treatment decision--a randomized trial among women with heavy menstruation. Health Expect. 2003 Dec;6(4):290-7. doi: 10.1046/j.1369-7625.2003.00225.x. PMID 15040791
- [Background] Dedianne MC, Hauzanneau P, Labarere J, Moreau A. Relation médecin-malade en soins primaires: qu'attendent les patients? Investigation par la méthode qualitative des focus groups. La revue du praticien Médecine générale. 2003;17 (612):653-6.
- [Background] Paul F, Jones MC, Hendry C, Adair PM. The quality of written information for parents regarding the management of a febrile convulsion: a randomized controlled trial. J Clin Nurs. 2007 Dec;16(12):2308-22. doi: 10.1111/j.1365-2702.2007.02019.x. PMID 18036121
- [Background] Sustersic M, Voorhoeve M, Menuret H, Baudrant M, Meneau A, Bosson JL. Fiches d'information pour les patients: quel intérêt? L'étude EDIMAP. La Revue de la médecine générale. 2010;276:332-9.
- [Background] Francis NA, Butler CC, Hood K, Simpson S, Wood F, Nuttall J. Effect of using an interactive booklet about childhood respiratory tract infections in primary care consultations on reconsulting and antibiotic prescribing: a cluster randomised controlled trial. BMJ. 2009 Jul 29;339:b2885. doi: 10.1136/bmj.b2885. PMID 19640941
- [Background] Lerman C, Ross E, Boyce A, Gorchov PM, McLaughlin R, Rimer B, Engstrom P. The impact of mailing psychoeducational materials to women with abnormal mammograms. Am J Public Health. 1992 May;82(5):729-30. doi: 10.2105/ajph.82.5.729. PMID 1566953
- [Result] Sustersic M, Meneau A, Dremont R, Paris A, Laborde L, Bosson JL. [Developing patient information sheets in general practice. Proposal for a methodology]. Rev Prat. 2008 Dec 15;58(19 Suppl):17-24. French. PMID 19253787
- [Result] Sustersic M, Meneau A, Dremont R, Bosson JL. Fiches d'information patient: quelle méthodologie? La revue du praticien Médecine générale. 2007;790:1167-8.
- [Result] Sustersic M, Meneau A, Drémont R, Paris A, Laborde L, Bosson JL. Elaboration d'un outil d'aide à l'éducation du patient pas la réalisation de 125 fiches d'information et de conseil concernant des motifs de consultation les plus fréquents en médecin générale. Université Joseph Fourier, faculté de médecine de Grenoble. juillet 2007.